CLINICAL TRIAL: NCT03561753
Title: Pilot Clinical Trial of PRS TB Regimen I - Phase II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Shanghai Center for Disease Control and Prevention (Other); No.85 Hospital, Changning, Shanghai, China (Other); Shanghai Public Health Clinical Center (Other Government); Bill and Melinda Gates Foundation (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Wei Sha MD & PhD, Director, Head of Tuberculosis Department,Shanghai Pulmonary Hospital, Principal Investigator, Clinical Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K18-103
Record Dates: First submitted 2018-05-21; First posted 2018-06-19 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Tuberculosis TB in Sputum: (+) Microscopy
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (the standard 2HRZE/4HR regimen) (Active Comparator): Group A, Standard Regimen (2EHRZ/4HR): Control group, use the standard six-month regimen with eight weeks of daily treatment with isoniazid, rifampin, ethambutol, and pyrazinamide followed by sixteen weeks of isoniazid and rifampin.
  Interventions: Drug: Group A (the standard 2HRZE/4HR regimen）
- Group B (New short course PRS regimen, 4EZ(high dose)PtoCfz) (Experimental): Group B, PRS Regimen (4EZ [high dose] Cfz Pto): Experience group，use the PRS regimen is 4 months of daily Cfz, Emb, Pto, and high dose pyrazinamide, dosed by weight.
  Interventions: Drug: Group B (New short course PRS regimen, 4EZ(high dose)PtoCfz)

INTERVENTIONS:
Drug: Group A (the standard 2HRZE/4HR regimen） — The standard six-month regimen is eight weeks of daily treatment with isoniazid, rifampin, ethambutol, and pyrazinamide followed by sixteen weeks of isoniazid and rifampin. The six-month regimen is the standard regimen for the treatment of drug-susceptible tuberculosis recommended by WHO.
  Other Names: The control group
  Arms: Group A (the standard 2HRZE/4HR regimen)
Drug: Group B (New short course PRS regimen, 4EZ(high dose)PtoCfz) — The PRS regimen I（new short course PRS regimen） is 4 months of daily Cfz, Emb, Pto, and high dose pyrazinamide, dosed by weight.Comparison of Standard Regimen：The standard six-month regimen is eight weeks of daily treatment with isoniazid, rifampin, ethambutol, and pyrazinamide followed by sixteen weeks of isoniazid and rifampin.
  Other Names: The experimental group
  Arms: Group B (New short course PRS regimen, 4EZ(high dose)PtoCfz)

SUMMARY:
Tuberculosis is the current leading cause of death due to an identifiable infectious agent worldwide. The current standard regimen for tuberculosis requires a patient to take drug combination (isoniazid, rifampicin, ethambutol, and pyrazinamide) for six to eight month periods. The purpose of this study is to compare tuberculosis treatment therapy between the current standard regimen and PRS derived combinatorial regimen. PRS derived regimen may potentially allow for a shorter course of treatment, which may reduce problems associated with adherence, toxicity, and development of drug resistance.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a major health problem of global proportions. Although drug sensitive TB is a treatable disease, the current standard treatment requires 6 - 8 months of a multi-drug regimen to achieve relapse-free cure. This long course of treatment is often associated with toxicity, poor compliance, and development of drug resistance. A more effective drug combination that provides more rapid sterilization of tissues has the potential to ameliorate these critical problems.

The current drug regimen for treating tuberculosis is lengthy and onerous, and hence complicated by poor compliance leading to drug resistance and disease relapse. Previously, using an output-driven optimization platform, parabolic response surface (PRS, previously called Feedback System control or FSC), and an in vitro macrophage model of Mycobacterium tuberculosis infection, we identified several new experimental drug regimens among billions of possible drug-dose combinations that outperform the current Standard Regimen. We used the PRS platform to optimize the in vivo drug doses of novel regimens (designated PRS regimen) in a mouse model of pulmonary tuberculosis and then showed that the regimens sterilized much more rapidly than the Standard Regimen and substantially reduced treatment time to relapse-free cure by 25% for PRS regimen, which consists of Clofazimine (Cfz), Ethambutol (E), high dose Pyrazinamide (Z, high), and Prothionamide (Pto). The regimen have the potential to provide a markedly shorter course of treatment for tuberculosis in humans. As PRS regimen omit isoniazid, rifampicin, fluoroquinolones, and injectable aminoglycosides, they are suitable for treating many cases of multidrug and extensively drug-resistant tuberculosis.

1 Significance of the study Based on results in cell culture in macrophages and in mice we anticipate that PRS regimen will prove to be more effective and will allow a shorter course of treatment than the standard regimen. By allowing a shorter course of treatment, problems with adherence, toxicity, and development of drug resistance can be reduced. Moreover, because the regimen does not include INH or RIF, it can be used in cases of TB that are resistant to those drugs.

2 Methods

1. Summary of Experimental Design This is a randomized, controlled, open-label pilot clinical trial. Previously untreated, smear positive tuberculosis patients (aged 18 - 65 years) with radiographic evidence of TB and whose bacteria are sensitive to first-line drugs will be randomly distributed to group A (standard regimen) and B (new short course PRS regimen). The study will compare sputum conversion rate at the end of treatment between treatment regimens and will evaluate objective indicators of treatment success rate and incidence of adverse events.
2. Identification of Subjects: Potentially eligible subjects will be identified from among subjects seen at or referred to the Shanghai Pulmonary Hospital for treatment of tuberculosis. Subjects will be informed about the study and those who express interest in participation will be provided a written consent form.
3. Consent Process: As described in detail below, Subjects will be informed that participation is voluntary and that they will receive appropriate care for their condition regardless of whether or not they participate in the study. Because subjects have active TB, they will be in isolation in the Shanghai Pulmonary Hospital. The investigator will review the consent form with the subject and ensure that the subject understands the consent form and that all of the subject's questions have been answered. Because timely initiation of treatment is important, subjects will be allowed up to two days to decide whether to participate in the study or to receive standard care.
4. Screening for Eligibility: Screening tests indicated in the Table of Study Procedures (located at the end of this document) and required for assessment of eligibility per inclusion/exclusion criteria will be completed within 14 days prior to study enrollment.
5. Randomization: Eligible subjects will be randomized 1:1 by using a random number generator either to Group A (standard care) or to Group B (the investigational PRS regimen).
6. Study Treatment: Subjects are treated according to their assignment to Group A or Group B as indicated below.

   Group A, Standard Regimen (2EHRZ/4HR): The standard six-month regimen is eight weeks of daily treatment with isoniazid, rifampin, ethambutol, and pyrazinamide followed by sixteen weeks of isoniazid and rifampin.

   All drugs are administered orally, seven days/week. Study drugs are dosed by weight as shown in the below. Group B, PRS Regimen (4EZ [high dose] Cfz Pto): The PRS regimen is 4 months of daily Cfz, Emb, Pto, and high dose pyrazinamide, dosed by weight according to below.

   The drug dosing for both Group A and Group B are summarized in the below:

   ………………………………………………………………………………………………………………………… Isoniazid (H):daily dose (gm)0.3(weight <50kg);0.3(weight≥50kg),use method: 1 times/day.

   Rifampin (R):daily dose (gm)0.45(weight <50kg);0.6(weight≥50kg),use method: 1 times/day（Fasting medication）.

   ethambutol (E):daily dose (gm)0.75(weight <50kg);1.0(weight≥50kg),use method: 1～2 times/day.

   pyrazinamide (Z):daily dose (gm)1.5(weight <50kg);1.5(weight≥50kg),use method:1～3 times/day.

   Pyrazinamide (High dose):daily dose (gm)1.75(weight <50kg);2.0(weight≥50kg),use method:1～2 times/day.

   clofazimine（Cfz）:daily dose (gm)0.15(weight <50kg);0.15(weight≥50kg),use method:1～3times/day.

   prothionamide（Pto）:daily dose (gm)0.6(weight <50kg);0.6(weight≥50kg),use method: 3 times/day.

   ……………………………………………………………………………………………………………
7. Patient follow up After 6-months standard treatment or 4-months short term PRS regimen treatment, subjects will have long term follow up to evaluate efficacy and ensure absence of relapse. The checkup times are at 1 month, 3 months, 6 months, 12 months and 24 months.

Evaluation of Efficacy i Bacteriology: sputum smear microscopy, culture using the Becton Dickinson Company mycobacterial growth indicator tube (MGIT) system and Lowenstein-Jensen (LJ) slant culture. MGIT testing will be used to evaluate drug susceptibility .

ii Radiology: All patients undergo chest X-ray and CT scan before treatment. X-ray will be reviewed after 8 weeks of treatment and at end of treatment and during the follow-up period. CT scan will be reviewed at end of treatment.

iii Bacterial load of sputum samples will be evaluated within two weeks after the start of treatment.

iv Time to culture positivity: Time to culture positivity will be performed by MGIT culture within two months after the start of treatment.

v Evaluation of results: We shall employ the World Health Organization (WHO) uniform standards in evaluating cure rate and treatment success rate, the sputum negative conversion rate, incidence of adverse events and patient compliance and other indicators. We shall compare these outcomes between the experimental group and the standard group to analyze the effect of each treatment regime.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed and untreated sputum smear positive tuberculosis patient
2. Pulmonary lesion consistent with TB by radiological examination
3. Positive sputum culture, identification of bacterial type confirmed Mycobacterium tuberculosis. MGIT drug sensitivity test (DST) results are sensitive of the first-line drugs (isoniazid, streptomycin, rifampicin and ethambutol).
4. Age 18 years-65 years old
5. Males or non-pregnant, non-nursing females
6. Women of child-bearing potential who are not surgically sterilized must agree to practice a barrier method of contraception or abstain from heterosexual intercourse during study drug treatment.

   a.Effective birth control methods: i.A double contraceptive method should be used as follows: ii.Double barrier method which can include any 2 of the following: a male condom, diaphragm, cervical cap, or female condom (male and female condoms should not be used together); or iii.Barrier method (one of the above) combined with hormone-based contraceptives or an intra-uterine device for the female subject/partner; iv.and are willing to continue practicing birth control methods throughout treatment and for 6 months (both male and female subjects) after the last dose of study medication or discontinuation from study medication in case of premature discontinuation.
7. Laboratory parameters done at or within 14 days prior to screening:

   1. Serum or plasma aminotransferases (AST, ALT) less than 3 times the upper limit of normal
   2. Serum or plasma total bilirubin less than or equal to 2.5 times the upper limit of normal
   3. Serum or plasma creatinine level less than or equal to 2 times the upper limit of normal
   4. Serum or plasma potassium level greater than or equal to 3.5 meq/L
   5. Hemoglobin level of 7.0 g/dL or greater
   6. Platelet count of 100,000/mm3 or greater
   7. For women of childbearing potential, a negative pregnancy test is required during screening
8. Provides written informed consent
9. Willingness and ability to attend scheduled follow-up visits and undergo study assessments.

Exclusion Criteria:

1. Tuberculosis resistant to any of the study drugs (isoniazid, rifampin, EMB, PZA, CFZ, Pto)
2. Unable to take oral medications.
3. History of allergy or intolerance to any of the study drugs
4. Serum aminotransferase (AST or ALT) 3x upper limit of normal or higher
5. Pregnant or nursing females, or plan to become pregnant or nurse during the study period
6. Males planning to conceive a child during the study or within 6 months of cessation of treatment.
7. Any treatment directed against active tuberculosis within 6 months preceding initiation of study drugs.
8. Suspected or documented tuberculosis involving the central nervous system and/or bones and/or joints, and/or miliary tuberculosis and/or pericardial tuberculosis.
9. HIV infected
10. HBV infected or HCV infected (these increase the risk of TB-drug induced hepatotoxicity)
11. Weight less than 40.0 kg.
12. Known allergy or intolerance to any of the study medications.
13. Individuals will be excluded from enrollment if, at the time of enrollment, their M. tuberculosis isolate is already known to be resistant to any of the study drugs.
14. QTcF > 500 msec
15. Other medical conditions, that, in the investigator's judgment, make study participation not in the individual's best interest.
16. Current or planned incarceration or other involuntary detention
17. Having participated in other clinical studies with dosing of investigational agents within 8 weeks prior to trial start or currently enrolled in an investigational study that includes treatment with medicinal agents. Subjects who are participating in observational studies or who are in a follow up period of a trial that included drug therapy may be considered for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
The rate of sputum smear/culture negative conversion | Group A (the standard 2HRZE/4HR regimen)：at the end of Sixth months after treatment. Group B (New short course PRS regimen, 4EZ(high dose)PtoCfz) ：at the end of Fourth months after treatment.
  The primary efficacy outcome is the proportion of the rate of sputum smear and culture(MGIT and LJ) negative conversion from samples collected at the end of treatment.

SECONDARY OUTCOMES:
Radiological manifestation change of lung TB lesions or cavity | Group A (the standard 2HRZE/4HR regimen)：at the end of Sixth months after treatment. Group B (New short course PRS regimen, 4EZ(high dose)PtoCfz) ：at the end of Fourth months after treatment.
  Radiological manifestation change of lung TB lesions or cavity at the end of treatment will be compared with those before treatment(Lesion size, absorption and improvement rate, and cavity closure rate, by chest x-ray and chest CT scans).
Number of Patients with Grade 3 or 4 Adverse Events | Group A (the standard 2HRZE/4HR regimen)：6 months from the beginning of clinical trials. Group B (New short course PRS regimen, 4EZ(high dose)PtoCfz) ：4 months from the beginning of clinical trials.
  Using a Modified Division of Acquired Immunodeficiency Syndrome National Institute of Allergy and Infectious Diseases [DAIDS] Scale of Adverse Event Reporting
Number of Patients with TB recurrence/relapse | 24 months after treatment completion for 2 groups.
  Number of Patients with TB recurrence/relapse by 24 months after the end of treatment(bacteriology and radiological examination confirmed).

CONTACTS AND LOCATIONS:
Overall Officials: sha wei, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (4):
- China (4):
  - Eighty-fifth Hospital of PLA, Shanghai
  - Shanghai Public Health Clinical Center Shanghai, China, Shanghai
  - Shanghai Center for Disease Control and Prevention, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai, China, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zumla A, Nahid P, Cole ST. Advances in the development of new tuberculosis drugs and treatment regimens. Nat Rev Drug Discov. 2013 May;12(5):388-404. doi: 10.1038/nrd4001. PMID 23629506
- [Background] Zumla A, Chakaya J, Centis R, D'Ambrosio L, Mwaba P, Bates M, Kapata N, Nyirenda T, Chanda D, Mfinanga S, Hoelscher M, Maeurer M, Migliori GB. Tuberculosis treatment and management--an update on treatment regimens, trials, new drugs, and adjunct therapies. Lancet Respir Med. 2015 Mar;3(3):220-34. doi: 10.1016/S2213-2600(15)00063-6. Epub 2015 Mar 9. PMID 25773212
- [Background] Nuermberger EL, Spigelman MK, Yew WW. Current development and future prospects in chemotherapy of tuberculosis. Respirology. 2010 Jul;15(5):764-78. doi: 10.1111/j.1440-1843.2010.01775.x. Epub 2010 Jun 4. PMID 20546189
- [Background] Ma Z, Lienhardt C, McIlleron H, Nunn AJ, Wang X. Global tuberculosis drug development pipeline: the need and the reality. Lancet. 2010 Jun 12;375(9731):2100-9. doi: 10.1016/S0140-6736(10)60359-9. Epub 2010 May 18. PMID 20488518
- [Background] Silva A, Lee BY, Clemens DL, Kee T, Ding X, Ho CM, Horwitz MA. Output-driven feedback system control platform optimizes combinatorial therapy of tuberculosis using a macrophage cell culture model. Proc Natl Acad Sci U S A. 2016 Apr 12;113(15):E2172-9. doi: 10.1073/pnas.1600812113. Epub 2016 Mar 28. PMID 27035987
- [Background] Lee BY, Clemens DL, Silva A, Dillon BJ, Maslesa-Galic S, Nava S, Ding X, Ho CM, Horwitz MA. Drug regimens identified and optimized by output-driven platform markedly reduce tuberculosis treatment time. Nat Commun. 2017 Jan 24;8:14183. doi: 10.1038/ncomms14183. PMID 28117835
- [Background] Handbook of anti-tuberculosis agents. Introduction. Tuberculosis (Edinb). 2008 Mar;88(2):85-6. doi: 10.1016/S1472-9792(08)70002-7. No abstract available. PMID 18486036
- [Background] Saukkonen JJ, Cohn DL, Jasmer RM, Schenker S, Jereb JA, Nolan CM, Peloquin CA, Gordin FM, Nunes D, Strader DB, Bernardo J, Venkataramanan R, Sterling TR; ATS (American Thoracic Society) Hepatotoxicity of Antituberculosis Therapy Subcommittee. An official ATS statement: hepatotoxicity of antituberculosis therapy. Am J Respir Crit Care Med. 2006 Oct 15;174(8):935-52. doi: 10.1164/rccm.200510-1666ST. PMID 17021358
- See also: WHO. 2015. Global Tuberculosis Report 2015. — http://www.who.int/tb/publications/global_report/en/